CLINICAL TRIAL: NCT06217029
Title: Applied Research on Young and Middle-aged Patients With Cervical Spondylotic Pain Using T2-mapping, T1ρ and Diffusion Kurtosis Imaging
Brief Title: Magnetic Resonance Imaging Study on Young and Middle-aged Patients With Cervical Spondylotic Pain
Acronym: MRI-CervPain
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2023-030
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain
Keywords: neck pain; young adults; T2-mapping; T1ρ; DKI
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities; Massage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Effective Group of Cervical Spondylotic Pain: VAS reduction rate is used to evaluate clinical efficacy. The reduction rate = (baseline value - end value)/baseline value. The clinical efficacy is divided into four levels: cured, significant effect, slight effect, ineffective or recurrent. cured: reduction rate ≥ 75%; significant effect: 50% ≤ reduction rate < 75%; slight effect: 25% ≤ reduction rate < 50%; ineffective: reduction rate < 25%. The "cured + significant effect" group was classified as the treatment effective group,
  Interventions: Other: physiotherapy and maxillary traction
- Ineffective Group of Cervical Spondylotic Pain: The "slight effect + ineffective" group and the recurrent group were classified as the treatment ineffective group
  Interventions: Other: physiotherapy and maxillary traction

INTERVENTIONS:
Other: physiotherapy and maxillary traction — 1. Mobility exercises
  2. Ultrasound or electric stimulation
  3. Application of equipment, such as braces, slings and taping
  4. Registered massage therapy
  5. Trigger point and myofascial release
  Other Names: massage therapy

SUMMARY:
Cervical and shoulder pain in young adults is commonly caused by intervertebral disc degeneration, bulge or herniation. Disc degeneration includes the synthetic and degradative imbalance of myxoid matrix, degeneration of annulus collagen, and decrease of water content in nucleus pulposus. A few patients with cervical degeneration had moderate to severe pain, but there are no obvious abnormalities in the shape and signal of the disc with routine MRI, which may be related to the early discal degeneration. In most cases, the pain could be relieved by non-surgical treatment due to mild decreased proteoglycan and slight abnormality of water diffusion, but these changes cannot be clearly demonstrated by routine MRI. Therefore, it is necessary to rely on sensitive MRI techniques to reflect the abnormal microstructure in the nucleus pulposus and annulus fibrosus, so as to assist the early detection of the main reason in patients with neck and shoulder pain and the evaluation of the efficacy of treatment.

DETAILED DESCRIPTION:
This is an observational, longitudinal, and single-center study. Confirmed patients with cervical and shoulder pain will complete several clinical and imaging programs before and after 3 and 12 months of non-surgical treatment for exploring the main reason of the symptom and the imaging predictors of treatment effect in the disease. The collected materials are listed below: (1) 3 times cervical MRI scans, including T2-mapping, T1ρ and DKI sequences, (2) visual analog scale (for pain assessment) and disease duration. Then the T2 value, T1ρ, and DKI derived parameters will be measured in the nucleus pulposus and annulus fibrosus.

ELIGIBILITY:
Inclusion Criteria:

1. Neck and shoulder pain, with or without upper limb pain and numbness;
2. Disease duration longer than 2 months
3. Visual analogue score (VAS) ≥ 3
4. Cervical MRI showing cervical disc degeneration, bulge, protrusion, etc.
5. Patients will undergo non-surgical treatment (maxillary occipital traction, massage, etc.)

Exclusion Criteria:

1. Severe trauma and surgery in neck and shoulder region.
2. X-ray or CT showing the severe cervical spine hyperplasia, infection (suppurative, tuberculous), neoplasm (various primary and secondary tumors), rheumatic (rheumatoid arthritis, ankylosing spondylitis), and nuclei pulposus calcification.
3. Cervical MRI revealed organic lesions such as inflammation of the spinal cord, tumors, syringomyelia, etc.
4. Chronic pain in other regions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults patients with neck and shoulder pain, who will undergo cervical spine MRI and non-surgical treatment
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
T1ρ alteration before and after 12 months treatment | 0, 12 months
  T1ρ imaging, which probes the interaction between water molecules and their macromolecular environment, has the potential to identify early biochemical changes in the intervertebral disc. There are correlations between T1ρ and glycosaminoglycan content, suggesting that T1ρ may be sensitive to early biochemical changes in disc degeneration. T1ρ will be measured in the nucleus pulposus, anterior and posterior annulus fibrosus of the cervical intervertebral disc.
Alterations of MK value before and after 12 months treatment | 0, 12 months
  Diffusion MRI techniques are noninvasive and quantitative techniques that can assess intervertebral disc degeneration by offering information about the properties of the water molecular diffusion process in intervertebral disc. In vivo tissues, the diffusion of water molecules has been hindered and restricted by complex microstructures, leading to a non-Gaussian probability distribution function. As a non-Gaussian model, diffusion kurtosis imaging (DKI) has a higher potential to characterize both molecular water diffusion and the complexity of tissue microstructures. DKI technique can provide several quantitative parameters, and the most important one is mean kurtosis (MK). MK value will be measured in the nucleus pulposus, anterior and posterior annulus fibrosus of the cervical intervertebral disc.

SECONDARY OUTCOMES:
T2* value alteration before and after 12 months treatment | 0, 12 months
  T2* mapping is sensitive to collagen fiber network. There is close correlation between T2* mapping and Pfirrmann grade, where a decrease in T2* value is significantly associated with the aggravation of intervertebral disc degeneration. Pathologically, T2* value is regarded as a robust biomarker at an earlier stage of disc degeneration. T2* value will be measured in the nucleus pulposus, anterior and posterior annulus fibrosus of the cervical intervertebral disc.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhang, M.D., Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhuang L, Wang L, Xu D, Wang Z, Liang R. Association between excessive smartphone use and cervical disc degeneration in young patients suffering from chronic neck pain. J Orthop Sci. 2021 Jan;26(1):110-115. doi: 10.1016/j.jos.2020.02.009. Epub 2020 Mar 20. PMID 32205018
- [Result] Chen C, Huang M, Han Z, Shao L, Xie Y, Wu J, Zhang Y, Xin H, Ren A, Guo Y, Wang D, He Q, Ruan D. Quantitative T2 magnetic resonance imaging compared to morphological grading of the early cervical intervertebral disc degeneration: an evaluation approach in asymptomatic young adults. PLoS One. 2014 Feb 3;9(2):e87856. doi: 10.1371/journal.pone.0087856. eCollection 2014. PMID 24498384
- [Result] Chen P, Wu C, Huang M, Jin G, Shi Q, Han Z, Chen C. Apparent Diffusion Coefficient of Diffusion-Weighted Imaging in Evaluation of Cervical Intervertebral Disc Degeneration: An Observational Study with 3.0 T Magnetic Resonance Imaging. Biomed Res Int. 2018 Feb 18;2018:6843053. doi: 10.1155/2018/6843053. eCollection 2018. PMID 29670903
- [Result] Leonova O, Baykov E, Sanginov A, Krutko A. Cervical Disc Degeneration and Vertebral Endplate Defects After the Fused Operation. Spine (Phila Pa 1976). 2021 Sep 15;46(18):1234-1240. doi: 10.1097/BRS.0000000000004007. PMID 33595261